CLINICAL TRIAL: NCT05724108
Title: A Phase II Randomized Control Trial of Triapine Plus Lutetium Lu 177 Dotatate Versus Lutetium Lu 177 Dotatate Alone for Well-Differentiated Somatostatin Receptor-Positive Neuroendocrine Tumors
Brief Title: Testing the Effectiveness of an Anti-cancer Drug, Triapine, When Used With Targeted Radiation-based Treatment (Lutetium Lu 177 Dotatate), Compared to Lutetium Lu 177 Dotatate Alone for Metastatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-01224; NCI-2023-01224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-CIRB-10558-PMC; 10558 (Other: Ohio State University Comprehensive Cancer Center LAO); 10558 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-02-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Specimen Handling; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (triapine, lutetium Lu 177 dotatate) (Experimental): Patients receive triapine PO QD on days 1-14 of each cycle and lutetium Lu 177 dotatate IV over 30 minutes on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Drug: Triapine
- Arm 2 (lutetium Lu 177 dotatate) (Active Comparator): Patients receive lutetium Lu 177 dotatate IV over 30 minutes on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Triapine — Given PO
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811
  Arms: Arm 1 (triapine, lutetium Lu 177 dotatate)

SUMMARY:
This phase II trial compares the effect of adding triapine to lutetium Lu 177 dotatate versus lutetium Lu 177 dotatate alone (standard therapy) in shrinking tumors or slowing tumor growth in patients with neuroendocrine tumors that have spread from where they first started (primary site) to other places in the body (metastatic). Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for deoxyribonucleic acid synthesis and cell growth. Lutetium Lu 177 dotatate is a radioactive drug. It binds to a protein called somatostatin receptor, which is found on some neuroendocrine tumor cells. Lutetium Lu 177 dotatate builds up in these cells and gives off radiation that may kill them. It is a type of radioconjugate and a type of somatostatin analog. Giving triapine in combination with lutetium Lu 177 dotatate may be more effective at shrinking tumors or slowing tumor growth in patients with metastatic neuroendocrine tumors than the standard therapy of lutetium Lu 177 dotatate alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of combination triapine + lutetium Lu 177 dotatate (treatment arm 1) versus standard of care lutetium Lu 177 dotatate alone (treatment arm 2).

SECONDARY OBJECTIVE:

I. Evaluate progression-free survival (PFS) between the two treatment arms (combination arm 1 versus standard of care arm 2).

EXPLORATORY OBJECTIVES:

I. Evaluate plasma hPG80 as a biomarker of treatment response. II. Evaluate plasma deoxyribonucleosides as a biomarker of triapine resistance. III. Collect plasma for circulating deoxyribonucleic acid (DNA) (ctDNA) assessment.

IV. Evaluate triapine plasma pharmacokinetics (PK) in the combination arm (treatment arm 1 only).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive triapine orally (PO) once daily (QD) on days 1-14 of each cycle and lutetium Lu 177 dotatate intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial.

ARM 2: Patients receive lutetium Lu 177 dotatate IV over 30 minutes on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 8 and 12 months, then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic, histologically confirmed well-differentiated neuroendocrine tumor with positive gallium 68 DOTATATE or copper 64 DOTATATE scan. Lesions on dotatate scan will be considered positive if the standardized uptake value maximum (SUVmax) of target lesion is > 2 times standardized uptake value (SUV) mean of normal liver parenchyma. Patients with lung neuroendocrine tumors (NETs) are excluded from the trial
* Patients must have progressive disease based on RECIST criteria, version 1.1 evidenced with CT scans/MRI obtained within 24 months from enrollment
* Patients must have measurable disease per RECIST 1.1
* Failure of at least one prior systemic cancer treatment with somatostatin analogs
* No prior exposure to peptide receptor radionuclide therapy
* Recovered from adverse events of previously administered therapeutic agents (i.e., to grade 2 or less toxicity) according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of triapine in combination with lutetium Lu 177 dotatate in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Serum creatinine =< 1.5 institutional ULN. Creatinine > 1.5 ULN will require a measured creatinine clearance (CrCl) > 50 ml/min to qualify
* Hemoglobin > 5.0 mmol/L (> 8.0 g/dL)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases and off steroids are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 4 weeks prior to enrollment in the study. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to enrollment in the study
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Pregnancy precaution: Men and women should avoid pregnancy for seven months after the date of their last treatment with lutetium Lu 177 dotatate. It is noteworthy that beta-human chorionic gonadotropin (beta-HCG) may be secreted by a small percentage of NETs, such that, in addition to being a pregnancy marker, it also is a tumor marker. Consequently, NET female patients with positive beta-HCG (> 5 mIU/mL) at baseline can be eligible to enter the study and receive treatment if pregnancy can be excluded by lack of expected doubling of beta-HCG and negative pelvic ultrasound. Normally, in pregnant subjects beta-HCG doubles every 2 days during the first 4 weeks of pregnancy and every 3.5 days by weeks 6 to 7. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months, and for women on hormone replacement therapy, only with a documented plasma follicle-stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral, implanted, or injected contraceptive hormones, an intrauterine device (IUD), or barrier methods (diaphragm, condoms, spermicidal) to prevent pregnancy, are practicing abstinence or where the partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential. Postmenopausal women who have fertilized eggs implanted are also considered to be of childbearing potential. Acceptable methods of contraception may include total abstinence at the discretion of the Investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensures compliance. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception (hormonal or barrier method of birth control; abstinence) should be maintained throughout the study and for 7 months after study treatment discontinuation. All men and women of childbearing potential and male partners must use a double-barrier method of birth control or practice continuous abstinence from heterosexual contact throughout the study and for seven months after the end of the last treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have not recovered from adverse events of previously administered therapeutic agents (i.e., have residual toxicities > grade 2) according to CTCAE 5.0, with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to triapine or lutetium Lu 177 dotatate
* Patients with uncontrolled intercurrent illness
* Uncontrolled congestive heart failure (New York Heart Association [NYHA] III, IV)
* Pregnant women are excluded from this study because triapine is a ribonucleotide reductase (RNR) inhibitor and lutetium Lu 177 dotatate is a peptide receptor radionuclide therapy with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with triapine and lutetium Lu 177 dotatate, breastfeeding should be discontinued if the mother is treated with triapine and lutetium Lu 177 dotatate and for 2.5 months following the last treatment
* Inability to swallow oral medications or gastrointestinal disease limiting absorption of oral agents
* Patients with any other significant condition, currently uncontrolled by treatment, which may interfere with completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 5 years
  Estimated along with exact 95% binomial confidence intervals in each arm and compared between arms using the z-test statistic.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from the date of randomization to the date of first documented progression or death due to any cause, assessed up to 5 years
  Progression will be measured by Response Evaluation Criteria in Solid Tumors 1.1 criteria. Log-rank test will be used to compare PFS between treatment and control. Median survival time and the corresponding confidence intervals will be calculated by the Kaplan-Meier Method.

OTHER OUTCOMES:
Plasma hPG80 | Up to 5 years
  Analysis of variance will be used to analyze plasma hPG80 concentration. Baseline plasma hPG80 will be used as covariate. F-test and t-test will be conducted to test the differences in hPG80 change between treatment arms and responses.
Plasma deoxyribonucleosides | Pre- to post-triapine administration
  Will evaluate plasma deoxyribonucleosides as a biomarker of triapine resistance. Pre and post triapine administration changes in deoxyribonucleosides will be analyzed by pair-wise t-test, stratified by study arm. Secondary and exploratory analysis on repeatedly measured deoxyribonucleosides will entail a linear mixed model for comparison between treatment groups.
Circulating deoxyribonucleic acid (ctDNA) | Up to 5 years
  ctDNA will be analyzed by summary descriptive statistics as well as visualization graphics such as heat maps. Data processing and downstream data analysis pipelines for the genomic data will be performed including differential analysis for comparison of genomic data between arms using the limma package in R/Bioconductor with adjustment for false discovery rate.
Triapine plasma pharmacokinetics (PK): Maximum concentration | Up to 5 years
  Will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated. PK parameters will be reported descriptively for exploratory comparison with historical data. Smoking status will be a particular covariate to be evaluated as a determinant of PK. Exploratory correlative studies with pharmacodynamics (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Triapine plasma PK: Area under the concentration-time curve | Up to 5 years
  Will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated. PK parameters will be reported descriptively for exploratory comparison with historical data. Smoking status will be a particular covariate to be evaluated as a determinant of PK. Exploratory correlative studies with pharmacodynamics (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Triapine plasma PK: Half-life | Up to 5 years
  Will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated. PK parameters will be reported descriptively for exploratory comparison with historical data. Smoking status will be a particular covariate to be evaluated as a determinant of PK. Exploratory correlative studies with pharmacodynamics (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Triapine plasma PK: Apparent clearance | Up to 5 years
  Will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated. PK parameters will be reported descriptively for exploratory comparison with historical data. Smoking status will be a particular covariate to be evaluated as a determinant of PK. Exploratory correlative studies with pharmacodynamics (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Triapine plasma PK: Apparent volume of distribution | Up to 5 years
  Will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated. PK parameters will be reported descriptively for exploratory comparison with historical data. Smoking status will be a particular covariate to be evaluated as a determinant of PK. Exploratory correlative studies with pharmacodynamics (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Lowell B Anthony, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (25):
- United States (25):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm